CLINICAL TRIAL: NCT01977924
Title: Impact of Polyphenols on Endothelial Function in Obstructive Sleep Apnea: a Randomized Controlled Trial
Brief Title: Impact of Polyphenols on Endothelial Function in Obstructive Sleep Apnea
Acronym: PolySAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-A00763-42
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea; polyphenols; endothelial function
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- polyphenols (Experimental): 600 mg polyphenols (grape extract)
  Interventions: Dietary Supplement: one month polyphenols supplementation (600mg)
- Placebo (Placebo Comparator): microcrystalline cellulose
  Interventions: Dietary Supplement: placebo (microcrystalline cellulose)

INTERVENTIONS:
Dietary Supplement: one month polyphenols supplementation (600mg)
  Arms: polyphenols
Dietary Supplement: placebo (microcrystalline cellulose)
  Arms: Placebo

SUMMARY:
Severe obstructive sleep apnea (OSA) is associated with increased cardiovascular morbidity and mortality. Endothelial dysfunction, an early marker of vascular disease has been demonstrated in OSA. Regular treatment of OSA by continuous positive airway pressure (CPAP) improves endothelial function and is associated with a reduction in cardiovascular risk. Approximately 40% of patients with OSA are intolerant or insufficiently adherent to CPAP. Alternative treatments or adjuvants to the CPAP are needed.

The polyphenols have demonstrated their effectiveness in improving endothelial function in patients with CV disease. No randomized controlled studies have evaluated the impact of PPR on the endothelial dysfunction associated with OSAHS.

DETAILED DESCRIPTION:
The endpoint is the change to one month of polyphenols treatment of the endothelial function measured by the index of hyperemic reactivity.

The secondary endpoints are changes at one month of supplementation with polyphenols of ambulatory blood pressure measurement in 24 hours (MAPA), micro-circulatory responsiveness, the speed of the pulse wave and biological measurements (lipid profile, blood glucose, fasting insulin, leptin, adiponectin, hs-CRP, 8-isoprostane levels and cellular origin of microparticles).

ELIGIBILITY:
Inclusion Criteria:•

* apnea hypopnea index > 30
* accepting polyphenols supplementation
* Signed informed consent

Exclusion Criteria:

* Epworth sleepiness scale > 16/24
* Severe cardiac and/or respiratory disease
* BMI>35 kg/m2
* Anemia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
endothelial function measured by the index of hyperemic reactivity | one month

REFERENCES:
- [Derived] Trzepizur W, Bironneau V, Recoquillon S, Priou P, Meslier N, Hamel JF, Henni S, Darsonval A, Messaoudi K, Martinez MC, Andriantsitohaina R, Gagnadoux F. Polyphenols Have No Impact on Endothelial Function in Patients with Obstructive Sleep Apnea: A Randomized Controlled Trial. J Nutr. 2018 Apr 1;148(4):581-586. doi: 10.1093/jn/nxy005. PMID 29659956